CLINICAL TRIAL: NCT02580305
Title: A Phase 2a Multicenter, Randomized, Double-Blind, Parallel Group, 26-Week, Placebo-Controlled Study of SUVN-502 in Subjects With Moderate Alzheimer's Disease Currently Treated With Donepezil Hydrochloride and Memantine Hydrochloride
Brief Title: SUVN-502 With Donepezil and Memantine for the Treatment of Moderate Alzheimer's Disease- Phase 2a Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suven Life Sciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTP2S1502HT6
Record Dates: First submitted 2015-10-17; First posted 2015-10-20 (Estimated); Results first posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Alzheimer's Disease
Keywords: SUVN-502; 5-HT6; Phase 2; Cognition; Donepezil; Memantine; Alzheimer's Disease; Triple Combination; Proof of Concept (POC)
MeSH Terms: conditions — Alzheimer Disease | interventions — 1-((2-bromophenyl)sulfonyl)-5-methoxy-3-((4-methyl-1-piperazinyl)methyl)-1H-indole dimesylate monohydrate; Donepezil; Namzaric; Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Experimental: SUVN-502 Low dose (50 mg) (Active Comparator): SUVN-502 Low dose adjunct to base treatment with Donepezil and Memantine
  Interventions: Drug: SUVN-502; Drug: Donepezil; Drug: Memantine
- Experimental: SUVN-502 High dose (100 mg) (Active Comparator): SUVN-502 High dose adjunct to base treatment with Donepezil and Memantine
  Interventions: Drug: SUVN-502; Drug: Donepezil; Drug: Memantine
- Placebo (Placebo Comparator): Placebo adjunct to base treatment with Donepezil and Memantine
  Interventions: Drug: Placebo; Drug: Donepezil; Drug: Memantine

INTERVENTIONS:
Drug: SUVN-502 — Once-daily, tablets, orally
  Other Names: Masupirdine
  Arms: Experimental: SUVN-502 High dose (100 mg); Experimental: SUVN-502 Low dose (50 mg)
Drug: Placebo — Once-daily, tablets, orally
  Arms: Placebo
Drug: Donepezil — Donepezil HCl (10 mg, once a day)
  Other Names: Namzaric
Drug: Memantine — Memantine HCl (10 mg, twice a day or 28 mg extended-release, once a day).
  Other Names: Namenda XR®

SUMMARY:
This is a phase 2a, proof-of-concept, 26-week, double-blind, multicenter, randomized, parallel group, placebo-controlled study to compare the efficacy and safety of treatment with SUVN-502 to placebo treatment in subjects with moderate Alzheimer's disease receiving stable doses of donepezil HCl and memantine HCl.

DETAILED DESCRIPTION:
This is a phase 2a, proof-of-concept, 26-week, double-blind, multicenter, randomized, parallel group, placebo-controlled study to compare the efficacy and safety of treatment with SUVN-502 to placebo treatment in subjects with moderate Alzheimer's disease receiving donepezil HCl (10 mg qd) and either memantine HCl (10 mg twice daily [bid]) or Namenda XR® (Extended Release, 28 mg qd) or the combination therapy, Namzaric™

The primary objective of the study is to evaluate the efficacy of a serotonin receptor subtype 6 (5-HT6) antagonist, SUVN-502, compared to placebo, as adjunct treatment in subjects with moderate Alzheimer's disease (Mini-Mental State Examination [MMSE] score of 12 to 20) currently treated with the acetylcholinesterase inhibitor, donepezil hydrochloride (HCl), and the N-methyl-D-aspartic acid (NMDA) antagonist, memantine HCl. Efficacy will be assessed by the 11-item Alzheimer's Disease Assessment Scale for Cognitive Behavior (ADAScog-11) after 26 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of probable Alzheimer's disease based on the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria at least 1 year prior to the screening visit.
* Has a score between 12 and 20 inclusive on the MMSE at the screening and baseline visits.
* Has a MRI or CT scan performed within 12 months prior to screening with findings consistent with the diagnosis of dementia due to Alzheimer's disease without any other clinically significant comorbid pathologies.
* Must be receiving treatment with stable doses of donepezil HCl and memantine HCl for at least 3 months prior to the screening visit
* Availability of an eligible and reliable caregiver
* Must be living in the community or an assisted living facility.
* Must be ambulatory or ambulatory aided (use of cane or walker).
* Is not pregnant or planning to become pregnant during the study.
* Subject (or subject's legally acceptable representative) and caregiver must sign an Informed Consent to participate in the study.

Exclusion Criteria:

* Has a diagnosis of dementia due to other than Alzheimer's Disease
* Is taking cholinesterase inhibitors other than donepezil HCl or taking doses of donepezil HCl other than 10 mg
* Is taking doses of memantine HCl other than 10 mg bid or Namenda XR® 28 mg qd.
* Has uncontrolled cardiac disease or hypertension.
* Has clinically significant renal or hepatic impairment.
* Has cancer or a malignant tumor, untreated thyroid disorder or has a history of seizure disorder
* Is treated or likely to require treatment during the study, with any medications prohibited by the study protocol.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2015-09; Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (71):
- United States (71):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Barrow Neurological Institute, Phoenix, Arizona
  - Territory Neurology & Research Institute, Tucson, Arizona
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Neuro-Pain Medical Center Inc, Fresno, California
  - Neurology Center of North Orange County, Fullerton, California
  - Senior Clinical Trials, Inc., Laguna Hills, California
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - Easton Center for Alzheimer's Disease Research at UCLA, Los Angeles, California
  - Paradigm Research, San Diego, California
  - Associated Neurologists of South Connecticut, Fairfield, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - Bradenton Research Center, Inc, Bradenton, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - CCM Clinical Research Group, Miami, Florida
  - Collier Neurologic Specialists, Naples, Florida
  - Palm Beach Neurological Center, Palm Beach Gardens, Florida
  - Anchor Neuroscience, Pensacola, Florida
  - Emerald Coast Center for Neurological Disorders, Pensacola, Florida
  - Neurostudies Inc, Port Charlotte, Florida
  - The Roskamp Institute, Inc., Sarasota, Florida
  - Brain Matters Research, Stuart, Florida
  - Neurology Clinical Research, Inc., Sunrise, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - University of South Florida - Byrd Alzheimer's Institute, Tampa, Florida
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Southern Illinois School of Medicine, Springfield, Illinois
  - Indiana University Health - University Hospital, Indianapolis, Indiana
  - Cotton-O'Neil Clinical Research Center, Topeka, Kansas
  - KU Medical Center Wichita Clinical Trial Unit, Wichita, Kansas
  - University Of Kentucky, Lexington, Kentucky
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Acadia Hospital, Bangor, Maine
  - Sheppard Pratt Health System, Baltimore, Maryland
  - Clinical Research Professionals, St Louis, Missouri
  - Princeton Medical Institute, Princeton, New Jersey
  - Advanced Memory Research Institute of NJ, PC - Internal Medicine, Rahway, New Jersey
  - Advanced Memory Research Institute, Toms River, New Jersey
  - Biobehavioral Health, Toms River, New Jersey
  - Neurology Specialists of Monmouth County, West Long Branch, New Jersey
  - Neurological Associates of Albany, PC, Albany, New York
  - Integrative Clinical Trials, LLC, Brooklyn, New York
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - Mid Hudson Medical Research, New Windsor, New York
  - New York University, New York, New York
  - Eastside Comprehensive Medical Center, LLC, New York, New York
  - Manhattan Behavioral Medicine, New York, New York
  - Upstate University Hospital (SUNY Health Science Center), Syracuse, New York
  - Five Towns Neuroscience Research, Woodmere, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - Alzheimer Memory Center, Charlotte, North Carolina
  - Richard Weisler, MD, PA, Raleigh, North Carolina
  - Ohio Clinical Research Partners, LLC, Canton, Ohio
  - Valley Medical Research, Centerville, Ohio
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Tulsa Clinical Research, LLC, Tulsa, Oklahoma
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Northeastern Pennsylvania Memory and Alzheimers Center, Plains, Pennsylvania
  - Roper St. Francis Healthcare, Charleston, South Carolina
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Shepherd Healthcare, Lewisville, Texas
  - Radiant Research, Inc., San Antonio, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Center for Alzheimer's Care, Imaging and Research, Salt Lake City, Utah
  - Independent Psychiatric Consultants, SC, dba, Waukesha, Wisconsin

REFERENCES:
- [Result] Nirogi R, Jayarajan P, Benade V, Shinde A, Goyal VK, Jetta S, Ravula J, Abraham R, Grandhi VR, Subramanian R, Pandey SK, Badange RK, Mohammed AR, Jasti V, Ballard C, Cummings J. Potential beneficial effects of masupirdine (SUVN-502) on agitation/aggression and psychosis in patients with moderate Alzheimer's disease: Exploratory post hoc analyses. Int J Geriatr Psychiatry. 2022 Oct;37(10):10.1002/gps.5813. doi: 10.1002/gps.5813. PMID 36168659
- [Result] Nirogi R, Ieni J, Goyal VK, Ravula J, Jetta S, Shinde A, Jayarajan P, Benade V, Palacharla VRC, Dogiparti DK, Jasti V, Atri A, Cummings J. Effect of masupirdine (SUVN-502) on cognition in patients with moderate Alzheimer's disease: A randomized, double-blind, phase 2, proof-of-concept study. Alzheimers Dement (N Y). 2022 Jun 1;8(1):e12307. doi: 10.1002/trc2.12307. eCollection 2022. PMID 35662833
- [Result] Nirogi R, Goyal VK, Benade V, Subramanian R, Ravula J, Jetta S, Shinde A, Pandey SK, Jayarajan P, Jasti V, Cummings J. Effect of Concurrent Use of Memantine on the Efficacy of Masupirdine (SUVN-502): A Post Hoc Analysis of a Phase 2 Randomized Placebo-Controlled Study. Neurol Ther. 2022 Dec;11(4):1583-1594. doi: 10.1007/s40120-022-00390-4. Epub 2022 Jul 31. PMID 35908254
- See also: Effect of Age, Cognitive Impairment Severity, and Duration of Disease on Efficacy of Masupirdine in Moderate Alzheimer's Disease Patients: A Post Hoc Analysis of a Phase-2 Randomized Placebo Controlled Study Results — https://doi.org/10.18103/mra.v10i9.3061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study centers located in the United States of America (USA) participated in the study
Groups:
- SUVN-502 Low Dose (50 mg): SUVN-502 Low dose (50 mg) adjunct to base treatment with Donepezil and Memantine
- SUVN-502 High Dose (100 mg): SUVN-502 High dose (100 mg) adjunct to base treatment with Donepezil and Memantine
Period: Overall Study
Arm/Group | SUVN-502 Low Dose (50 mg) | SUVN-502 High Dose (100 mg) | Placebo
Started | 190 | 185 | 189
Safety Population | 187 | 181 | 188
Modified Intent-to-treat (mITT) Population | 184 | 176 | 183
Completed | 147 | 136 | 157
Not Completed | 43 | 49 | 32
Not completed — Adverse Event | 15 | 19 | 10
Not completed — Lack of Efficacy | 5 | 0 | 2
Not completed — Protocol Violation | 4 | 9 | 6
Not completed — Lost to Follow-up | 4 | 4 | 2
Not completed — Withdrawal by Subject | 11 | 9 | 7
Not completed — Randomized in error and never treated | 4 | 8 | 5

BASELINE CHARACTERISTICS:
Population: A total of 564 patients were randomized as per the planned ratio to receive masupirdine 50 mg (190 patients), masupirdine 100 mg (185 patients), or placebo (189 patients). A total of 543 (96.3%) patients who were randomized to specific treatment sequence were included in the modified intent to treat (mITT) population and this mITT population is considered for baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | SUVN-502 Low Dose (50 mg) | SUVN-502 High Dose (100 mg) | Placebo | Total
Number analyzed (Participants) | 184 | 176 | 183 | 543
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.4 (8.08) | 74.4 (6.97) | 72.9 (7.23) | 73.6 (7.46)
Age, Customized [Count of Participants; unit: Participants]
  Age group greater than or equal to 65 years | 159 | 155 | 157 | 471
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 96 | 106 | 297
  Male | 89 | 80 | 77 | 246
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 3
  Asian | 3 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 6 | 8 | 10 | 24
  White | 171 | 162 | 168 | 501
  More than one race | 3 | 2 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
APO-E4 Carrier Status [Count of Participants; unit: Participants]
  Carrier one allele | 77 | 79 | 84 | 240
  Carrier two allele | 24 | 31 | 35 | 90
Mini-Mental State Examination [Mean (Standard Deviation); unit: units on a scale] — Mini-Mental State Examination (MMSE) was used to measure cognitive impairment. The MMSE can evaluate overall cognitive function, and is widely used for the assessment of cognitive impairment in dementia patients. The questionnaire consists of 11 items, and each item aims to evaluate different cognitive domains such as orientation, memory, attention, and construction. The score ranged from 0 to 30, with a higher score indicating better function.
  units on a scale | 16.9 (2.21) | 17.0 (2.47) | 16.5 (2.48) | 16.8 (2.39)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week-26 in Alzheimer's Disease Assessment Scale-Cognitive Subscale 11 (ADAS-Cog 11)
Description: Mean change from baseline at week 26 is assessed for ADAS-Cog11 score. The ADAS-Cog11 is a structured scale that evaluates memory, orientation, attention, reasoning, language, and constructional praxis. ADAS-Cog11 measures cognition by assessing 11 metrics impaired in AD: word recall; commands; constructional praxis; naming objects and fingers; ideational praxis; orientation; word recognition; remembering test instructions; spoken language ability; word-finding difficulty; and comprehension of spoken language. The scale ranges from 0 to 70, with higher scores indicate greater impairment.
Time Frame: Baseline to Week 26
Population: modified intent to treat (mITT) population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SUVN-502 Low Dose (50 mg) | SUVN-502 High Dose (100 mg) | Placebo
Number analyzed (Participants) | 184 | 176 | 183
score on a scale | 2.0 (0.5) | 2.5 (0.5) | 2.6 (0.5)
Statistical Analysis 1: Comparison: SUVN-502 Low Dose (50 mg) vs Placebo; Test type: Superiority; p = 0.41, Mixed Models Analysis — Threshold for statistical significance was p≤0.05; Statistical Method: Mixed model for repeated measures
Statistical Analysis 2: Comparison: SUVN-502 High Dose (100 mg) vs Placebo; Test type: Superiority; p = 0.90, Mixed Models Analysis — Threshold for statistical significance was p≤0.05; Statistical Method: Mixed model for repeated measures

2. Secondary Outcome: Change From Baseline to Week-26 in Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB)
Description: Clinical Dementia Rating-Sum of Boxes (CDR-SB) - Sum of Boxes CDR-SB is a semi-structured interview of participants and their caregivers. Participant's cognitive status is rated across 6 domains of functioning, including memory, orientation, judgment/problem solving, community affairs, home/hobbies, and personal care.
  Severity score assigned for each of 6 domains; total score (SB) ranges from 0 to 18. Higher scores indicate greater disease severity.
Time Frame: Baseline to Week 26
Population: modified intent to treat (mITT) population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SUVN-502 Low Dose (50 mg) | SUVN-502 High Dose (100 mg) | Placebo
Number analyzed (Participants) | 184 | 176 | 183
score on a scale | 1.3 (0.2) | 1.0 (0.2) | 1.2 (0.2)
Statistical Analysis 1: Comparison: SUVN-502 Low Dose (50 mg) vs Placebo; Test type: Superiority; p = 0.46, Mixed Models Analysis — Threshold for statistical significance was p≤0.05; Statistical Method: Mixed model for repeated measures
Statistical Analysis 2: Comparison: SUVN-502 High Dose (100 mg) vs Placebo; Test type: Superiority; p = 0.48, Mixed Models Analysis — Threshold for statistical significance was p≤0.05; Statistical Method: Mixed model for repeated measures

3. Secondary Outcome: Change From Baseline to Week-26 in Alzheimer's Disease Cooperative Study Group-Activities of Daily Living (ADCS-ADL)
Description: The Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL) Inventory Score is a 23-item inventory.
  The ADCS-ADL measures both basic and instrumental activities of daily living The total ADCS-ADL score ranges from 0 to 78, with lower scores indicating greater disease severity.
Time Frame: Baseline to Week 26
Population: modified intent to treat (mITT) population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SUVN-502 Low Dose (50 mg) | SUVN-502 High Dose (100 mg) | Placebo
Number analyzed (Participants) | 184 | 176 | 183
score on a scale | -4.6 (0.6) | -3.4 (0.6) | -4.4 (0.6)
Statistical Analysis 1: Comparison: SUVN-502 Low Dose (50 mg) vs Placebo; Test type: Superiority; p = 0.83, Mixed Models Analysis — Threshold for statistical significance was p≤0.05; Statistical Method: Mixed model for repeated measures
Statistical Analysis 2: Comparison: SUVN-502 High Dose (100 mg) vs Placebo; Test type: Superiority; p = 0.24, Mixed Models Analysis — Threshold for statistical significance was p≤0.05; Statistical Method: Mixed model for repeated measures

4. Secondary Outcome: Change From Baseline to Week-26 in Neuropsychiatric Inventory (NPI)
Description: Neuropsychiatric Inventory (NPI) 12 item - Total Score NPI assesses psychopathology in participants with dementia and other neurologic disorders.
  Total score ranges from 12 to 144; higher scores indicate greater disease severity.
Time Frame: Baseline to Week 26
Population: modified intent to treat (mITT) population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SUVN-502 Low Dose (50 mg) | SUVN-502 High Dose (100 mg) | Placebo
Number analyzed (Participants) | 184 | 176 | 183
score on a scale | 0.5 (0.8) | 0.4 (0.9) | 2.1 (0.8)
Statistical Analysis 1: Comparison: SUVN-502 Low Dose (50 mg) vs Placebo; Test type: Superiority; p = 0.17, Mixed Models Analysis — Threshold for statistical significance was p≤0.05; Statistical Method: Mixed model for repeated measures
Statistical Analysis 2: Comparison: SUVN-502 High Dose (100 mg) vs Placebo; Test type: Superiority; p = 0.14, Mixed Models Analysis — Threshold for statistical significance was p≤0.05; Statistical Method: Mixed model for repeated measures

5. Secondary Outcome: Change From Baseline to Week-26 in Change in Mini Mental State Examination (MMSE)
Description: Change in Mini-Mental State Examination (MMSE) - Total Score Minimum Score - 0, Maximum Score - 30. Higher score means better outcome.
Time Frame: Baseline to Week 26
Population: modified intent to treat (mITT) population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SUVN-502 Low Dose (50 mg) | SUVN-502 High Dose (100 mg) | Placebo
Number analyzed (Participants) | 184 | 176 | 183
score on a scale | -1.1 (0.3) | -1.1 (0.3) | -1.0 (0.3)
Statistical Analysis 1: Comparison: SUVN-502 Low Dose (50 mg) vs Placebo; Test type: Superiority; p = 0.79, Mixed Models Analysis — Threshold for statistical significance was p≤0.05; Statistical Method: Mixed model for repeated measures
Statistical Analysis 2: Comparison: SUVN-502 High Dose (100 mg) vs Placebo; Test type: Superiority; p = 0.92, Mixed Models Analysis — Threshold for statistical significance was p≤0.05; Statistical Method: Mixed model for repeated measures

ADVERSE EVENTS:
Time Frame: 26 Weeks
Description: Safety population is considered for reporting total number of participants at risk.
Arm/Group | SUVN-502 Low Dose (50 mg) | SUVN-502 High Dose (100 mg) | Placebo
All-Cause Mortality (participants affected / at risk) | 3/187 | 2/181 | 1/188
Serious Adverse Events (participants affected / at risk) | 10/187 | 14/181 | 12/188
Other Adverse Events (participants affected / at risk) | 50/187 | 44/181 | 40/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SUVN-502 Low Dose (50 mg) (N=187) | SUVN-502 High Dose (100 mg) (N=181) | Placebo (N=188)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SUVN-502 Low Dose (50 mg) (N=187) | SUVN-502 High Dose (100 mg) (N=181) | Placebo (N=188)
Urinary tract infection (Infections and infestations) | 15 (16) | 21 (26) | 19 (22)
Headache (Nervous system disorders) | 12 (12) | 4 (4) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 12 (14) | 9 (9) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 11 (16) | 10 (12) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-03-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT02580305/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/05/NCT02580305/SAP_001.pdf